CLINICAL TRIAL: NCT05810818
Title: Effectiveness Of Dry Needling and Soft Tissue Mobilization Combined With Self-Stretching for Management of Calf and Heel Pain
Brief Title: Effectiveness Of DN and STM Combined With Self-Stretching for Management of Calf and Heel Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/520
Record Dates: First submitted 2023-03-15; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Heel Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling along stretches and soft tissues therapy (Experimental)
  Interventions: Diagnostic Test: Dry Needling
- stretching and soft tissue mobilization (Active Comparator)
  Interventions: Diagnostic Test: Self Stretching

INTERVENTIONS:
Diagnostic Test: Dry Needling — Dry needling treatment will be consisting of two treatments per week
  Arms: Dry needling along stretches and soft tissues therapy
Diagnostic Test: Self Stretching — Self stretching groups both will receive a TrP manual interventions and stretching protocol
  Arms: stretching and soft tissue mobilization

SUMMARY:
To determine the effectiveness of dry needling and soft tissue mobilization with self-stretching for the management of calf and heel pain. In our topic pain and physical dysfunction are our variables

ELIGIBILITY:
Inclusion Criteria:

* Patients will be between the ages of 25 to 60 years.
* Female and males.
* History of heel and calf pain.
* Pain level moderate .
* Trigger point / inactive trigger points.
* Acute stage patients.

Exclusion Criteria:

* Phobias like injections or needles.
* Unwilling patients
* Patients on anticoagulant medicines.
* Patients with RA
* Fibromyalgia syndrome.
* Pateint with recent trauma and surgery.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Dry Needling and Soft Tissue Mobilization with Self-Stretching | 6 Months
  Effectiveness Of Dry Needling and Soft Tissue Mobilization Combined with Self-Stretching for Management of Calf and Heel Pain

IPD SHARING:
Plan to Share IPD: No